CLINICAL TRIAL: NCT06313450
Title: De-escalated Radiotherapy for Primary Tumor After Neoadjuvant Therapy With Toripalimab Plus Chemotherapy for Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Fang-Yun Xie, professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: B2023-110-X02
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Nasopharyngeal Carcinoma; Radiotherapy; Complications; IMMUNOTHERAPY
Keywords: Nasopharyngeal Carcinoma; de-escalated radiotherapy; immunotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- de-escalated radiotherapy (Experimental): If the primary tumour regresses by over 75% and the level of EBV DNA reduces to zero, a radiation dose of 60Gy will be administered. Additionally, three cycles of Toripalimab (240mg, every three weeks) and two cycles of cisplatin (100mg/m2, every three weeks) will be given during radiotherapy.
  Interventions: Radiation: de-escalated radiotherapy
- conventional radiotherapy (Other): If the primary tumour regresses by less than 75% or if EBV DNA remains above zero, a conventional radiation dose of 70Gy to the primary tumor and two cycles of cisplatin (100mg/m2, every three weeks) will be administered during radiotherapy.
  Interventions: Radiation: conventional radiotherapy

INTERVENTIONS:
Radiation: de-escalated radiotherapy — Enrolled patients receive three courses of induction therapy with gemcitabine and cisplatin, along with Toripalimab. After induction therapy, patients with a tumor volume regression of 75% or more and no detectable EBV DNA will receive de-escalated radiotherapy for the primary tumor with 60 Gy. During radiotherapy, patients will receive Cisplatin 100 mg/m2 every three weeks for two courses and Toripalimab 240 mg every three weeks for three courses. If patients do not achieve complete remission at the end of radiotherapy, 6 Gy will be added to the residual lesions.
  Arms: de-escalated radiotherapy
Radiation: conventional radiotherapy — Enrolled patients receive three courses of induction therapy with gemcitabine and cisplatin, along with Toripalimab. After induction therapy, patients with tumor volume regression less than 75% or EBV DNA copy number higher than 0 receive conventional radiotherapy for the primary tumor with 70 Gy. Patients will receive Cisplatin 100 mg/m2, every three weeks for two courses during radiotherapy.
  Arms: conventional radiotherapy

SUMMARY:
In the IMRT era, patients with stage II-III (AJCC8th) nasopharyngeal carcinoma achieve high local control. However, survivors are increasingly experiencing late radiation-induced toxicities. A previous study found that reducing the radiation dose to the primary site to 60Gy for patients who achieved partial or complete response to induction chemotherapy resulted in a lower rate of late toxicities and an inferior local control rate. The investigators aim to reduce the radiation dose to the primary site for patients after immunochemotherapy, given the potential of neoadjuvant chemotherapy and immunotherapy to increase response rates and long-term survival. The protocol includes participants with stage II-III (AJCC8th), except T2N0M0, to receive three courses of neoadjuvant gemcitabine plus cisplatin and Toripalimab. If the primary tumour regresses by over 75%, de-escalated radiotherapy with 60Gy will be administered, and participants will receive two cycles of cisplatin and three cycles of Toripalimab during the radiotherapy course. Otherwise, participants will receive conventional radiotherapy and concurrent chemotherapy with cisplatin for two cycles as usual. The aim of this study is to investigate the 3-year local control rate and toxicities of de-escalated radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed nasopharyngeal carcinoma, patients who have not received anti-cancer therapy;
2. ECOG performance status score (PS score) 0 or 1.
3. 18-70 years old.
4. Stage II-III except T2N0M0 (AJCC 8th).
5. Neutrophil count ≥ 1.5 × 10^9/L, hemoglobin ≥ 90 g/L and platelet count ≥ 100 × 10^9/L.
6. Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≤ 2.5 times the upper limit of normal (ULN), bilirubin ≤ 1.5 times ULN; Creatinine clearance ≥ 60 ml/min
7. Patients are required to sign an informed consent form and must be willing and able to comply with the visits, treatment plan, laboratory tests, and other requirements specified in the study protocol

Exclusion Criteria:

Patients will be excluded from the study, if any of the following criteria is met:

1. Over the age of 70 or under the age of 18.
2. HBsAg positive and HBV DNA ≥ 1 × 10^3 copies/ml
3. HCV antibody positive.
4. Subjects with active, known or suspected autoimmune diseases were excluded from the study. Eligible participants included those with type 1 diabetes mellitus, hypothyroidism requiring only hormone replacement therapy, and skin conditions that do not require systemic therapy such as vitiligo, psoriasis, or alopecia.
5. History of interstitial lung disease;
6. Receiving systemic sex hormones or other immunosuppressive therapy at equivalent doses ≥ 10 mg prednisone/day within 28 days prior to signing informed consent; Subjects with systemic sex hormone doses ≤ 10 mg prednisone/day or inhaled/topical corticosteroids were eligible.
7. Received or about to receive live vaccines within 30 days before signing the informed consent form;
8. Pregnant or lactating women;
9. Other malignancies within 5 years, except carcinoma in situ, adequately treated non-melanoma skin cancer and papillary thyroid cancer;
10. Known previous hypersensitivity to macromolecular protein preparations, or to any component of Toripalimab;
11. Human immunodeficiency virus (HIV) infection.
12. Other conditions that may affect the safety of subjects or trial compliance as judged by the investigator, including symptomatic heart failure, unstable angina pectoris, myocardial infarction, active infection requiring systemic treatment, mental illness or family and social factors;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 112 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
local recurrence rate(LRR) | 3 years
  Defined as the proportion of patients with local recurrence within 3 years

SECONDARY OUTCOMES:
primary tumor volume regression≥75% rate | Two weeks after the third cycle of neoadjuvant immunochemotherapy (each cycle is 21 days), prior to radiotherapy
3-year overall survival | 3 years
acute and late radiation-induced toxicities | up to 3 years after radiotherapy, respectively
complete response rate of primary tumor | Two weeks after the third cycle of neoadjuvant immunochemotherapy (each cycle is 21 days) and six months after radiotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] undefined
- [Result] Liu YP, Wen YH, Tang J, Wei Y, You R, Zhu XL, Li J, Chen L, Ling L, Zhang N, Zou X, Hua YJ, Chen YM, Chen L, Lu LX, Chen MY, Wen WP. Endoscopic surgery compared with intensity-modulated radiotherapy in resectable locally recurrent nasopharyngeal carcinoma: a multicentre, open-label, randomised, controlled, phase 3 trial. Lancet Oncol. 2021 Mar;22(3):381-390. doi: 10.1016/S1470-2045(20)30673-2. Epub 2021 Feb 15. PMID 33600761
- [Result] Peng H, Chen L, Zhang Y, Li WF, Mao YP, Liu X, Zhang F, Guo R, Liu LZ, Tian L, Lin AH, Sun Y, Ma J. The Tumour Response to Induction Chemotherapy has Prognostic Value for Long-Term Survival Outcomes after Intensity-Modulated Radiation Therapy in Nasopharyngeal Carcinoma. Sci Rep. 2016 Apr 21;6:24835. doi: 10.1038/srep24835. PMID 27099096
- [Result] Yao JJ, Jin YN, Lin YJ, Zhang WJ, Marks T, Ryan I, Zhang HY, Xia LP. The feasibility of reduced-dose radiotherapy in childhood nasopharyngeal carcinoma with favorable response to neoadjuvant chemotherapy. Radiother Oncol. 2023 Jan;178:109414. doi: 10.1016/j.radonc.2022.11.003. Epub 2022 Nov 11. PMID 36375563
- [Result] Chen AM, Felix C, Wang PC, Hsu S, Basehart V, Garst J, Beron P, Wong D, Rosove MH, Rao S, Melanson H, Kim E, Palmer D, Qi L, Kelly K, Steinberg ML, Kupelian PA, Daly ME. Reduced-dose radiotherapy for human papillomavirus-associated squamous-cell carcinoma of the oropharynx: a single-arm, phase 2 study. Lancet Oncol. 2017 Jun;18(6):803-811. doi: 10.1016/S1470-2045(17)30246-2. Epub 2017 Apr 20. PMID 28434660
- [Result] Marur S, Li S, Cmelak AJ, Gillison ML, Zhao WJ, Ferris RL, Westra WH, Gilbert J, Bauman JE, Wagner LI, Trevarthen DR, Balkrishna J, Murphy BA, Agrawal N, Colevas AD, Chung CH, Burtness B. E1308: Phase II Trial of Induction Chemotherapy Followed by Reduced-Dose Radiation and Weekly Cetuximab in Patients With HPV-Associated Resectable Squamous Cell Carcinoma of the Oropharynx- ECOG-ACRIN Cancer Research Group. J Clin Oncol. 2017 Feb 10;35(5):490-497. doi: 10.1200/JCO.2016.68.3300. Epub 2016 Dec 28. PMID 28029303
- [Result] OuYang PY, Zhang BY, Guo JG, Liu JN, Li J, Peng QH, Yang SS, He Y, Liu ZQ, Zhao YN, Li A, Wu YS, Hu XF, Chen C, Han F, You KY, Xie FY. Deep learning-based precise prediction and early detection of radiation-induced temporal lobe injury for nasopharyngeal carcinoma. EClinicalMedicine. 2023 Apr 4;58:101930. doi: 10.1016/j.eclinm.2023.101930. eCollection 2023 Apr. PMID 37090437
- [Result] Tang LL, Guo R, Zhang N, Deng B, Chen L, Cheng ZB, Huang J, Hu WH, Huang SH, Luo WJ, Liang JH, Zheng YM, Zhang F, Mao YP, Li WF, Zhou GQ, Liu X, Chen YP, Xu C, Lin L, Liu Q, Du XJ, Zhang Y, Sun Y, Ma J. Effect of Radiotherapy Alone vs Radiotherapy With Concurrent Chemoradiotherapy on Survival Without Disease Relapse in Patients With Low-risk Nasopharyngeal Carcinoma: A Randomized Clinical Trial. JAMA. 2022 Aug 23;328(8):728-736. doi: 10.1001/jama.2022.13997. PMID 35997729
- [Result] Zhang Y, Chen L, Hu GQ, Zhang N, Zhu XD, Yang KY, Jin F, Shi M, Chen YP, Hu WH, Cheng ZB, Wang SY, Tian Y, Wang XC, Sun Y, Li JG, Li WF, Li YH, Mao YP, Zhou GQ, Sun R, Liu X, Guo R, Long GX, Liang SQ, Li L, Huang J, Long JH, Zang J, Liu QD, Zou L, Su QF, Zheng BM, Xiao Y, Guo Y, Han F, Mo HY, Lv JW, Du XJ, Xu C, Liu N, Li YQ, Xie FY, Sun Y, Ma J, Tang LL. Final Overall Survival Analysis of Gemcitabine and Cisplatin Induction Chemotherapy in Nasopharyngeal Carcinoma: A Multicenter, Randomized Phase III Trial. J Clin Oncol. 2022 Aug 1;40(22):2420-2425. doi: 10.1200/JCO.22.00327. Epub 2022 Jun 16. PMID 35709465